CLINICAL TRIAL: NCT06566651
Title: Emotion and Interoception Processing in ALS
Brief Title: Emotion Processing Among Patients With ALS
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mia Heintzelmann, Ph.d. fellow, University of Aarhus
Other Study IDs: emotionperceptionALS11072308
Record Dates: First submitted 2023-11-28; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; ALS; Motor Neuron Disease; MND (Motor Neurone DIsease)
Keywords: Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Emotion Perception; Emotion Processing; Emotion Recognition; Autonomic Responses; Respiratory Responses; Heart rate; Emotion Discrimination Task; ALS; Motorneuron disease; MND
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amyotrophic Lateral Sclerosis (ALS): People diagnosed or suspected of having the neurodegenerative disease Amyotrophic Lateral Sclerosis (ALS)
  Interventions: Other: Emotion Discrimination Task (EDT)
- Neuromuscular: People diagnosed with a neuromuscular disease other than ALS
  Interventions: Other: Emotion Discrimination Task (EDT)
- Control: Healthy people
  Interventions: Other: Emotion Discrimination Task (EDT)

INTERVENTIONS:
Other: Emotion Discrimination Task (EDT) — It estimates the subjective bias and sensitivity in discriminating between happy and angry facial expressions of different intensities of emotional expression

SUMMARY:
The goal of this observational study is to learn about the emotional perception in people with ALS disease compared to people with other neuromuscular disease and healthy controls. The main questions it aims to answer are:

* How people with ALS judge happy and angry faces and what their "insight" into these judgements are like
* How their autonomic responses differ from the other two test group Participants will asked to judge if a face presents a happy emotion or angry emotion.

Researchers will compare the ALS group responses with neuromuscular diseases group and healthy control group responses to see if the ALS group judge more happy faces than angry.

DETAILED DESCRIPTION:
Mild cognitive and behavioral changes occur in 35% of ALS patients and 10-15% of patients meet the criteria for FTD1-4. Recent research suggests changes in emotional perception and social cognition are a part of the neuropsychological changes in ALS, possibly associated with cognitive and behavioral symptoms seen in ALS-FTD5-9.

The aim of this project is to investigate emotional perception in ALS patients compared to healthy controls and patients with other neuromuscular diseases that do not affect the central nervous system. We use a simple emotion discrimination task to evaluate emotional bias and metacognition of emotion discrimination. Moreover, this project aims to explore the correlation between emotion perception and autonomic reactivity in ALS patients by recording heart rate frequency and respiration frequency during the EDT.

The project will contribute with deeper insights to the neuropsychological changes in ALS patients and the opportunity to quantify these changes. Thereby, the project will add new perspectives to the discussion of how we evaluate socio-emotional aspects of ALS in both clinical decision-making, guidance of relatives and future research.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients, ambulant and hospitalized

  * Able to give informed consent
  * Diagnosed with ALS or probable ALS according to the existing revision of the El Escorial Criteria 21,22.
* Patients with a peripheral neuromuscular disease, ambulant and hospitalized

  * Able to give informed consent
  * Diagnosed with a peripheral neuromuscular disease, that does not affect CNS, including but not limited to Myasthenia Gravis and polyneuropathy
* Healthy controls

  * Able to give informed consent
  * Age and gender matched to ALS patients

Exclusion Criteria:

* All Participants

  * Other severe medical, neurological, or psychiatric disorders
  * Visual impairment to an extent that interferes with the ability to perform of the test
  * Severe motor or cognitive deficits, to the extent that the test-task cannot be performed
  * Alcohol or drug abuse to an extent the interferes with task performance
* Patients with a peripheral neuromuscular disease

  ● Familial predisposition to ALS
* Healthy controls

  * Familial predisposition to ALS (first degree relatives)
  * Medical treatment that affects the central nervous system (e.g., antidepressants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Residents of Aarhus and Aalborg
  * Patients at Aarhus University Hospital
  * Patients at Aalborg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The perception of facial emotions measured using an Emotion Discrimination Task (EDT). | 20 minutes
  The EDT requires subjects to assess the facial emotion of a face stimulus and report whether the facial emotion was angry or happy. This will be the operationalisation of subjects' emotion perception, which we anticipate will reveal a bias towards positive perceptions. There is thus two scores on this scale: "Angry" and "Happy". There is no one of these scores that is "better" than the other. It is an nominal categorical scare.
Metacognitive sensitivity measured using a retrospective confidence rating scale | 20 minutes
  Metacognitive insight will be operationalized through a metacognitive sensitivity measure. The method employed for this is a confidence rating measure, where subjects assess their own performance on the EDT. Subjects will indicate on a sliding scale, ranging from "very confident" (maximum score) to a "pure guess" (minimum score), how confident they are that their previous answer was correct. Generally higher scores on this scale is considered better. This scales title is: " Confidence Rating Scale".

SECONDARY OUTCOMES:
Subjects' heart rate is monitored throughout the EDT | 20 minutes
  Subjects heart rate is measured through a standard 3-lead electrocardiogram montage. Electrodes were place on both collarbones and on the left lower rib.
Subjects' respiration is monitored throughout the EDT | 20 minutes
  Subjects' respiration is measured using a respiratory belt around the upper torso.

CONTACTS AND LOCATIONS:
Overall Officials: Mia B Heintzelmann, Cand.med, Principal Investigator — Department of Neurology, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Aalborg University Hospital, Aalborg, Region Nordjulland

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD. Once the data is fully anonymized, they may be released on public scientific repositories such as Github or Figshare.
Time Frame: After the anonymizing the data, which is set to happen after collecting the data from the last participant being tested, the data will become available. The data will be available for minimum of 3 years.
Access Criteria: Through approval by Aarhus University Hospital or Region Midtjylland can individuals receive the collected data. The data can potentially be used as part of a masters thesis.

REFERENCES:
- [Background] Swinnen B, Robberecht W. The phenotypic variability of amyotrophic lateral sclerosis. Nat Rev Neurol. 2014 Nov;10(11):661-70. doi: 10.1038/nrneurol.2014.184. Epub 2014 Oct 14. PMID 25311585
- [Background] Sedda A. Disorders of emotional processing in amyotrophic lateral sclerosis. Curr Opin Neurol. 2014 Dec;27(6):659-65. doi: 10.1097/WCO.0000000000000147. PMID 25333604
- [Background] Strong MJ, Abrahams S, Goldstein LH, Woolley S, Mclaughlin P, Snowden J, Mioshi E, Roberts-South A, Benatar M, HortobaGyi T, Rosenfeld J, Silani V, Ince PG, Turner MR. Amyotrophic lateral sclerosis - frontotemporal spectrum disorder (ALS-FTSD): Revised diagnostic criteria. Amyotroph Lateral Scler Frontotemporal Degener. 2017 May;18(3-4):153-174. doi: 10.1080/21678421.2016.1267768. Epub 2017 Jan 5. PMID 28054827
- [Background] Strong MJ, Yang W. The frontotemporal syndromes of ALS. Clinicopathological correlates. J Mol Neurosci. 2011 Nov;45(3):648-55. doi: 10.1007/s12031-011-9609-0. Epub 2011 Aug 2. PMID 21809041
- [Background] Bora E. Meta-analysis of social cognition in amyotrophic lateral sclerosis. Cortex. 2017 Mar;88:1-7. doi: 10.1016/j.cortex.2016.11.012. Epub 2016 Dec 5. PMID 28002755
- [Background] Martins AP, Prado LGR, Lillo P, Mioshi E, Teixeira AL, de Souza LC. Deficits in Emotion Recognition as Markers of Frontal Behavioral Dysfunction in Amyotrophic Lateral Sclerosis. J Neuropsychiatry Clin Neurosci. 2019 Spring;31(2):165-169. doi: 10.1176/appi.neuropsych.18040086. Epub 2018 Dec 12. PMID 30537912
- [Background] Oh SI, Oh KW, Kim HJ, Park JS, Kim SH. Impaired Perception of Emotional Expression in Amyotrophic Lateral Sclerosis. J Clin Neurol. 2016 Jul;12(3):295-300. doi: 10.3988/jcn.2016.12.3.295. Epub 2016 Apr 19. PMID 27095526
- [Background] Zimmerman EK, Eslinger PJ, Simmons Z, Barrett AM. Emotional perception deficits in amyotrophic lateral sclerosis. Cogn Behav Neurol. 2007 Jun;20(2):79-82. doi: 10.1097/WNN.0b013e31804c700b. PMID 17558250
- [Background] Lule D, Kurt A, Jurgens R, Kassubek J, Diekmann V, Kraft E, Neumann N, Ludolph AC, Birbaumer N, Anders S. Emotional responding in amyotrophic lateral sclerosis. J Neurol. 2005 Dec;252(12):1517-24. doi: 10.1007/s00415-005-0907-8. Epub 2005 Jun 24. PMID 15977000
- [Background] Crespi C, Cerami C, Dodich A, Canessa N, Arpone M, Iannaccone S, Corbo M, Lunetta C, Scola E, Falini A, Cappa SF. Microstructural white matter correlates of emotion recognition impairment in Amyotrophic Lateral Sclerosis. Cortex. 2014 Apr;53:1-8. doi: 10.1016/j.cortex.2014.01.002. Epub 2014 Jan 18. PMID 24534360
- [Background] Lule D, Diekmann V, Anders S, Kassubek J, Kubler A, Ludolph AC, Birbaumer N. Brain responses to emotional stimuli in patients with amyotrophic lateral sclerosis (ALS). J Neurol. 2007 Apr;254(4):519-27. doi: 10.1007/s00415-006-0409-3. Epub 2007 Mar 31. PMID 17401515
- [Background] Aho-Ozhan HE, Keller J, Heimrath J, Uttner I, Kassubek J, Birbaumer N, Ludolph AC, Lule D. Perception of Emotional Facial Expressions in Amyotrophic Lateral Sclerosis (ALS) at Behavioural and Brain Metabolic Level. PLoS One. 2016 Oct 14;11(10):e0164655. doi: 10.1371/journal.pone.0164655. eCollection 2016. PMID 27741285
- [Background] Finegan E, Chipika RH, Li Hi Shing S, Hardiman O, Bede P. Pathological Crying and Laughing in Motor Neuron Disease: Pathobiology, Screening, Intervention. Front Neurol. 2019 Mar 21;10:260. doi: 10.3389/fneur.2019.00260. eCollection 2019. PMID 30949121
- [Background] Caga J, Hsieh S, Lillo P, Dudley K, Mioshi E. The Impact of Cognitive and Behavioral Symptoms on ALS Patients and Their Caregivers. Front Neurol. 2019 Mar 11;10:192. doi: 10.3389/fneur.2019.00192. eCollection 2019. PMID 30915018
- [Background] de Wit J, Bakker LA, van Groenestijn AC, van den Berg LH, Schroder CD, Visser-Meily JMA, Beelen A. Caregiver burden in amyotrophic lateral sclerosis: A systematic review. Palliat Med. 2018 Jan;32(1):231-245. doi: 10.1177/0269216317709965. Epub 2017 Jul 3. PMID 28671483
- [Background] Olney RK, Murphy J, Forshew D, Garwood E, Miller BL, Langmore S, Kohn MA, Lomen-Hoerth C. The effects of executive and behavioral dysfunction on the course of ALS. Neurology. 2005 Dec 13;65(11):1774-7. doi: 10.1212/01.wnl.0000188759.87240.8b. PMID 16344521
- [Background] Borasio GD, Miller RG. Clinical characteristics and management of ALS. Semin Neurol. 2001 Jun;21(2):155-66. doi: 10.1055/s-2001-15268. PMID 11442324
- [Background] Benbrika S, Desgranges B, Eustache F, Viader F. Cognitive, Emotional and Psychological Manifestations in Amyotrophic Lateral Sclerosis at Baseline and Overtime: A Review. Front Neurosci. 2019 Sep 10;13:951. doi: 10.3389/fnins.2019.00951. eCollection 2019. PMID 31551700
- [Background] Lule D, Ehlich B, Lang D, Sorg S, Heimrath J, Kubler A, Birbaumer N, Ludolph AC. Quality of life in fatal disease: the flawed judgement of the social environment. J Neurol. 2013 Nov;260(11):2836-43. doi: 10.1007/s00415-013-7068-y. Epub 2013 Aug 30. PMID 23989341
- [Background] Garcia-Cordero I, Migeot J, Fittipaldi S, Aquino A, Campo CG, Garcia A, Ibanez A. Metacognition of emotion recognition across neurodegenerative diseases. Cortex. 2021 Apr;137:93-107. doi: 10.1016/j.cortex.2020.12.023. Epub 2021 Jan 28. PMID 33609899
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Wang S, Adolphs R. Reduced specificity in emotion judgment in people with autism spectrum disorder. Neuropsychologia. 2017 May;99:286-295. doi: 10.1016/j.neuropsychologia.2017.03.024. Epub 2017 Mar 24. PMID 28343960